CLINICAL TRIAL: NCT05552118
Title: A Post-Market, Prospective, Multi-Centre, Open-Label, Comparative, Interventional Study of Adult Cochlear Implant Speech Performance and Clinic Efficiency With Remote Care (Remote Check & Remote Assist) Compared With Standard of Care in the First 12 Months Post-initial Activation
Brief Title: Speech Performance and Clinic Efficiency With Remote Care Compared With Standard of Care in Adults With a Cochlear Implant in the First 12 Months Post-activation
Acronym: INSPIRE
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cochlear (Industry)
Collaborators: QbD Clinical (Industry); Avania (Industry); TFS (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: CLTD5764
Record Dates: First submitted 2022-09-06; First posted 2022-09-23 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2025-09

CONDITIONS: Hearing Loss
Keywords: Cochlear Implant aftercare; Remote clinical management
MeSH Terms: conditions — Hearing Loss | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cochlear™ Remote care (Experimental): Is composed of Cochlear™ Remote Check and Cochlear™ Remote Assist.
  Interventions: Procedure: Cochlear™ Remote care; Device: Compatible Implant Series and Compatible Sound Processors
- Standard of care (Active Comparator): Routine In-clinic care
  Interventions: Procedure: Standard of care; Device: Compatible Implant Series and Compatible Sound Processors

INTERVENTIONS:
Procedure: Cochlear™ Remote care — Cochlear™ Remote Check is a virtual assessment tool which helps the clinician to monitor the participant hearing progress remotely. It allows the participant to complete a series of hearing tests using the Cochlear™ Nucleus® Smart App then electronically send the results to the clinician for review.
  Cochlear™ Remote Assist enables a video call appointment through the Cochlear™ Custom Sound® Pro software and the Nucleus® Smart App. When remote check requires further follow-up, it allows the clinician to make programming adjustments and sound processor settings without a clinic visit.
  Arms: Cochlear™ Remote care
Procedure: Standard of care — Routine in clinic face-to-face care and sound processor programming using Cochlear™ Custom Sound® Pro
  Arms: Standard of care
Device: Compatible Implant Series and Compatible Sound Processors — Individuals who are implanted with a compatible cochlear implant series and compatible sound processor are eligible to participate.

SUMMARY:
The aim of the study is to assess the real-world effectiveness of managing participants within the first year post-activation (between 3 and 12 months) using Cochlear's Remote Care (Remote Check and Remote Assist), as compared with standard in-clinic management. The study captures also the time and costs associated with both models of care to quantify the potential costs savings and efficiency gains possible with delivering Cochlear Implant (CI) aftercare remotely.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years or older (no upper age limit)
* Post-lingually deafened or pre-lingually deafened with measurable word scores in quiet using a cochlear implant
* Unilaterally implanted with a compatible Cochlear™ implant
* Currently using a compatible Cochlear™ Sound Processor
* 3 months, +/- 2 weeks, experience with a cochlear implant (post-activation) at the time of baseline measurements
* Direct access to a compatible Smart Phone
* Fluent in the languages used for the study, as determined by the investigator
* Willing to participate in and comply with all requirements of the protocol, including willingness to be randomised to either arm
* Willing and able to provide written informed consent

Exclusion Criteria:

* Patient has a MAP incompatible with Master Volume, Bass and Treble (MVBT) programming:

  * Non-monopolar MAPs (bipolar, common ground, variable mode)
  * Dynamic range of <10 Comfortable Level (CL)
  * Hybrid mode enabled
  * Pulse widths >100 µs
  * 10 or more electrodes turned off
* Patient has on-going fluctuations in MAP Threshold levels (Ts) and Comfort levels (Cs) and/or impedances
* Patient requires frequent individual channel measurements and/or measurements without the use of live-stimulation
* Score below 3 on the screening subset of questions from the Mobile Device Proficiency Questionnaire (MDPQ)
* Abnormal cochlea anatomy and/or facial nerve stimulation that requires complex or more frequent programming, as determined by the Investigator
* Additional disabilities that would prevent participation in evaluations, including significant visual impairment and/or dexterity issues
* Unable or unwilling to comply with the requirements of the clinical investigation as determined by the Investigator
* Investigator site personnel directly affiliated with this study and/or their immediate families; immediate family is defined as a spouse, parent, child, or sibling
* Cochlear employees or employees of Contract Research Organisations or contractors engaged by Cochlear for the purposes of this investigation
* Current participation, or participation in another interventional clinical study/trial in the past 30 days, involving an investigational drug or device (unless the other investigation was/is a Cochlear sponsored investigation and determined by the investigator or Sponsor to not impact this investigation).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 148 (Estimated)
Dates: Start 2024-03-18 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Mean change in patient reported hearing ability in daily life measured with the SSQ12 (Speech, Spatial and Qualities of Hearing Scale) questionnaire between month 3 (baseline) and month 12 post-activation | 3 months post-activation (baseline) and 12 months post-activation
  Measuring change of speech, spatial and hearing experiences (12 items). Each item is scored on a scale of 0 to 10 where 0 corresponds to "complete inability or complete absence of a quality" and 10 to "complete ability or complete presence of an ability". The score of a participant is determined as the mean of the 12 items. Higher scores indicate less hearing disability

SECONDARY OUTCOMES:
Mean change in speech recognition score for an open-set word recognition measure in quiet between 3 months post-activation (baseline) and 12 months post-activation | 3 months post-activation (baseline) and 12 months post-activation
  The test is done using phonetically balanced words and scores are recorded as % correct words. Higher scores indicate a better outcome.
Mean change in speech recognition score for sentences in adaptive noise between 3 months post-activation (baseline) and 12 months post-activation | 3 months post-activation (baseline) and 12 months post-activation
  The test is done using validated lists of phonetically balanced sentences. The noise is kept constant at 65 decibel (dB) Sound Pressure Level (SPL), and the speech is adapted stepwise to establish the speech-to-noise ratio (SNR) providing a 50% level of understanding. Lower scores indicate a better outcome.
Descriptive summaries of clinic time and resource utilisation incurred between 3 months and 12 months post-activation assessed via a custom questionnaire. | 3 months post-activation (baseline) and 12 months post-activation
Descriptive summaries of time and costs incurred by participants between 3 months and 12 months post-activation via a custom questionnaire | 3 months post-activation (baseline) and 12 months post-activation
Participant satisfaction measured with the Client Satisfaction Questionnaire (CSQ)-8 at 12 months post-activation | 12 months post-activation
  Measuring satisfaction of participants with the healthcare service (8 questions). Each item is scored using a 4-point Likert scale with 1 always indicating a negative response and 4 a positive response. A total higher score indicates higher satisfaction
Participant empowerment measured with the Patient Activation Measure (PAM), at 12 months post-activation | 12 months post-activation
  Evaluating the knowledge, skills, beliefs, and behaviours that participants have for self-management of their long-term health condition (13 items). Each item is scored on a 4-point likert scale from 1 (strongly disagree) to 4 (strongly agree). The overall score is calculated and normalized to a 100-point scale. Higher scores indicate greater levels of activation.

CONTACTS AND LOCATIONS:
Overall Officials: Katie Keyrouse, Study Director — Cochlear
Locations (11):
- Ear Science Institute Australia, Subiaco, Western Australia, Australia
- Belgium (2):
  - UZ Gent, Ghent
  - UZ Leuven, Leuven
- Italy (2):
  - University of Bari "A. Moro" UOC Otorinolaringoiatria Universitaria, Bari
  - Azienda Ospedale Università di Padova, Padua
- Netherlands (2):
  - Academisch Ziekenhuis Maastricht, Maastricht
  - Radboud University Medical Centre Nijmegen, Nijmegen
- United Kingdom (4):
  - Queen Elizabeth Hospital Audiology Centre - University Hospital Birmingham, Birmingham
  - Auditory Implant Centre, Glan Clwyd Hospital, Bodelwyddan
  - St Thomas' Hospital, London
  - St George's Hospital, London

IPD SHARING:
Plan to Share IPD: No
Cochlear do not have an approved platform for public sharing of IPD collected in this study. Data may be provided to individual researchers on request.

REFERENCES:
- [Derived] Quaranta N, Murri A, Denys S, Verhaert N, Huinck W, Townsend J, Swinnen F, Dhooge I, de Klerk A, Mehta D, Brotto D, Craddock L, Hoskam G, Schou IM, McBride ME, Campbell-Bell C. Randomised controlled trial to assess the efficiency and effectiveness of remote care compared with in-clinic care for adult cochlear implant recipients in the first 12 months after activation: a protocol of the INSPIRE study. BMJ Open. 2025 Oct 20;15(10):e094283. doi: 10.1136/bmjopen-2024-094283. PMID 41120152